CLINICAL TRIAL: NCT03942107
Title: The Effect of Dental Post Application After Root Canal Treatment on Postoperative Pain in Asymptomatic Teeth.
Brief Title: Postoperative Pain After Dental Post Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Tan Firat Eyuboglu, Assistant Professor, Head of Department of Endodontics, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: dental posts postop pain
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Pain; Endodontically Treated Teeth; Vibration; Exposure
Keywords: Dental posts; postoperative pain; single-visit root canal treatment; two-visit root canal treatment; vibration
MeSH Terms: conditions — Pain, Postoperative; Tooth, Nonvital

STUDY DESIGN:
Intervention Model Description: after root canal treatment, post and core application in the first group and only root canal treatment in the second group post operative pain intensity will be assessed at 24, 48, and 72-h; 7-day follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: RCT+post+core in 1 visit (Active Comparator): the root canal treatment will be completed with 2Shape NiTi system as well as post and core application in the same visit prior to postoperative pain evaluation.
  Interventions: Procedure: Group 1: single-visit RCT
- Group 2: after RCT, post and core in 2nd visit (Active Comparator): after root canal treatment conducted with 2Shape NiTi system, the postoperative pain evaluation will be completed prior applying post and core for coronal restoration.
  Interventions: Procedure: Group 2: two-visit RCT

INTERVENTIONS:
Procedure: Group 1: single-visit RCT — both root canal treatment and post and core restoration of the coronal part of the tooth is completed in single visit prior to postoperative pain evaluation at 24, 48 and 72-h and 7-day follow-up time
  Other Names: 1-visit RCT
  Arms: Group 1: RCT+post+core in 1 visit
Procedure: Group 2: two-visit RCT — after root canal treatment is completed, postoperative pain evaluation will be conducted in this group at 24, 48 and 72-h and 7-day follow-up time. post-core application will be completed at the seventh day after postoperative pain evaluation.
  Other Names: 2-visit RCT
  Arms: Group 2: after RCT, post and core in 2nd visit

SUMMARY:
In this study the effect of dental post application on postoperative dental pain in patients with asymptomatic teeth after a single-appointment root canal treatment will be evaluated.

DETAILED DESCRIPTION:
The aim of this clinical study is to evaluate the effect of dental post application on postoperative pain intensity level in patients with asymptomatic teeth after a single-appointment root canal treatment. A total of one hundred patients with asymptomatic teeth and with no contradictory medical history who are indicated for non-surgical root canal treatment and application of a dental post at the Endodontic Clinic, Faculty of Dentistry, Istanbul Medipol University, between April and December of 2019 will be included. All of the patients will be recruited from the Istanbul Medipol University Dental Clinics in Istanbul. the patients will be divided in two groups (n=50). Consent will be obtained from all study participants before the treatment. After the root canal treatments are completed in single-visit, in the first groups dental posts will be applied immediately at the same visit and patients will be appointed for pain assessment. In group 2 after the root canal treatment a temporary filling be applied in the access cavity and patients will be appointed for pain assessment. Dental posts will be applied after the pain assessment is completed at the end of 1 week. All treatments will be performed by one endodontist. Postoperative pain intensity will be assessed at 24, 48, and 72 h; 7 days; after the treatment. The teeth will be examined according to postoperative pain intensity levels,

ELIGIBILITY:
Inclusion Criteria:

* patients with asymptomatic teeth which were in need of orthograde non-surgical root canal treatment with post application

Exclusion Criteria:

Patients

* who were younger than 18 years old,
* who had contradictory medical history for root canal treatment,
* who used antibiotics 1 month prior and analgesics 1 week prior to the treatment,
* who could not abide the follow-up time Teeth
* that were symptomatic
* with previous root canal treatment
* with present or suspected vertical root fracture
* with ≥ 4 mm periodontal pocket depth
* with apical lesions ≥ 5mm
* with damaged or resorbed apex
* that were in need of apical surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Postoperative Pain after post and core application in root canal traeted teeth | 24, 48, and 72 hours; 7 days
  The primary outcome measure of the study is to assess if the application of post and core to restore coronal part of root canal treated teeth may have an additive effect on postoperative pain intensity. Postoperative pain is recorded using vertical Visual Analog Scale (VAS) at 24, 48, and 72-h and 7-day follow-up time by one operator. Patients are asked to mark their pain level on a vertical line with the end points "No pain" and "Worst possible pain". The distance of the marked point to "no pain" end point is measured to calculated pain intensity level. The longer the distance the more the pain intensity level is.

CONTACTS AND LOCATIONS:
Overall Officials: TAN F EYUBOGLU, DDS,PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University School of Dentistry, Istanbul, Turkey (Türkiye)